CLINICAL TRIAL: NCT00706238
Title: Study of GSK1203486A Antigen-Specific Cancer Immunotherapeutic in Patients With Unresectable and Progressive Metastatic Cutaneous Melanoma
Brief Title: MAGE-A3 Antigen-Specific Cancer Immunotherapeutic in Patients With Progressive Metastatic Cutaneous Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to difficulties in recruiting subjects, not following concerns for the safety or absence of clinical activity in patients.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110551; 2007-005203-18 (EudraCT Number)
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Melanoma
Keywords: metastatic,; Melanoma,; Antigen-Specific Cancer Immunotherapeutic,; ASCI; MAGE-A3; tumor antigen,
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis

ARMS (1):
- GSK1203486A Group (Experimental): Patients received 4 cycles of MAGE-A3 product as follows:
  * Cycle 1: 6 doses, each given at a 2-week interval,
  * Cycle 2: 6 doses, each given at a 3-week interval
  * Cycle 3: 4 doses, each given at a 6-week interval
  * Cycle 4: 4 doses, each given at a 3-month interval followed by 4 doses, each given at a 6-month interval.
  The MAGE-A3 product was administered intramuscularly in the deltoid or lateral regions of the thighs, alternately on the right and left sides.
  Interventions: Biological: GSK Biologicals' Recombinant MAGE-A3 Antigen-Specific Cancer Immunotherapeutic (ASCI) GSK1203486A

INTERVENTIONS:
Biological: GSK Biologicals' Recombinant MAGE-A3 Antigen-Specific Cancer Immunotherapeutic (ASCI) GSK1203486A — IM administration in the deltoid or lateral regions of the thighs, alternately on the right and left sides.

SUMMARY:
This study is being done to evaluate the safety and the clinical activity of MAGE-A3 Antigen-Specific Cancer Immunotherapeutic in patients with unresectable and progressive metastatic cutaneous melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient with histologically proven, measurable metastatic cutaneous melanoma, and with documented progressive disease within the 12 weeks before the first administration of study treatment.
* Written informed consent has been obtained from the patient before the performance of any protocol-specific procedure.
* Patient is >= 18 years of age at the time of signature of the informed consent.
* The patient's tumor shows expression of MAGE-A3 gene
* ECOG performance status of 0 or 1.
* The patient has normal organ functions
* If the patient is female, she must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to administration of study treatment, have a negative pregnancy test and continue such precautions during all study treatment period and for 2 months after completion of the injection series.
* In the view of the investigator, the patient can and will comply with the requirements of the protocol.

Exclusion Criteria:

* The patient has at any time received systemic (bio-)chemotherapy (except for isolated limb perfusion, as long as this was performed at least 4 weeks before first study treatment administration).
* The patient is scheduled to receive any anti-cancer specific treatment, including radiotherapy, immunotherapy, chemotherapy and immunomodulating agents.
* The patient requires concomitant treatment with systemic corticosteroids, or any other immunosuppressive agents.
* The patient received any cancer immunotherapeutic containing a MAGE-A3 antigen or any cancer immunotherapeutic for his/her metastatic disease.
* The patient has received any investigational or non-registered drug or vaccine other than the study medication within the 30 days preceding the first ASCI injection or it is planned that (s)he will receive such a drug during the study period.
* The patient has (or has had) previous or concomitant malignancies at other sites, except effectively treated malignancy that is considered by the investigator highly likely to have been cured.
* History of allergic disease or reactions likely to be exacerbated by any component of the study investigational product.
* The patient has an autoimmune disease such as, but not limited to, multiple sclerosis, lupus, and inflammatory bowel disease. Patients with vitiligo are not excluded.
* The patient has a family history of congenital or hereditary immunodeficiency.
* The patient is known to be positive for the Human Immunodeficiency Virus (HIV).
* The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent, or to comply with the trial procedures.
* The patient has concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
* For female patients: the patient is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-09-29 (Actual); Primary Completion 2011-01-19 (Actual); Study Completion 2011-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Argentina (3):
  - GSK Investigational Site, CABA, Buenos Aires
  - GSK Investigational Site, Quilmes, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
- GSK Investigational Site, Athens, Greece
- GSK Investigational Site, Oslo, Norway

RESULTS

PARTICIPANT FLOW:
Groups:
- GSK1203486A Group: Patients received 4 cycles of MAGE-A3 product as follows: - Cycle 1: 6 doses, each given at a 2-week interval, - Cycle 2: 6 doses, each given at a 3-week interval - Cycle 3: 4 doses, each given at a 6-week interval - Cycle 4: 4 doses, each given at a 3-month interval followed by 4 doses, each given at a 6-month interval. The MAGE-A3 product was administered intramuscularly in the deltoid or lateral regions of the thighs, alternately on the right and left sides.
Period: Overall Study
Arm/Group | GSK1203486A Group
Started | 5
Completed | 0
Not Completed | 5
Not completed — Disease progression | 4
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | GSK1203486A Group
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Antigen-Specific Cancer Immunotherapeutic (ASCI) Related Grade 3/4 Adverse Events (AE)
Description: The assessment was made as per the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, where Grade refers to the severity of the AE. The CTCAE version 3.0 displays Grades 1 through 5 with unique clinical descriptions of severity for each AE, as follows: Grade 1 = Mild AE; Grade 2 = Moderate AE; Grade 3 = Severe AE; Grade 4 = Life-threatening or disabling AE; Grade 5 = Death related to AE.
Time Frame: During the entire study, up to 2.5 years per patient
Population: The Total treated cohort (TTC) included all patients who received at least one dose of the ASCI.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1203486A Group
Number analyzed (Participants) | 5
Participants | 0

2. Primary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study, up to 2.5 years per patient
Population: The Total treated cohort (TTC) included all patients who received at least one dose of the ASCI.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1203486A Group
Number analyzed (Participants) | 5
Participants | 1

3. Primary Outcome: The Rate of Objective Clinical Response.
Time Frame: At the time of analysis.
Population: As the study was terminated before the end of recruitment, data was not collected.
Arm/Group | GSK1203486A Group
Number analyzed (Participants) | 0

4. Secondary Outcome: The Rate of Stable Disease.
Time Frame: At the time of analysis.
Population: As the study was terminated before the end of recruitment, data was not collected.
Arm/Group | GSK1203486A Group
Number analyzed (Participants) | 0

5. Secondary Outcome: The Rate of Mixed Response.
Time Frame: At the time of analysis.
Population: As the study was terminated before the end of recruitment, data was not collected.
Arm/Group | GSK1203486A Group
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Study Treatment Failure.
Time Frame: At the time of analysis.
Population: As the study was terminated before the end of recruitment, data was not collected.
Arm/Group | GSK1203486A Group
Number analyzed (Participants) | 0

7. Secondary Outcome: Progression-free Survival.
Time Frame: At the time of analysis.
Population: As the study was terminated before the end of recruitment, data was not collected.
Arm/Group | GSK1203486A Group
Number analyzed (Participants) | 0

8. Secondary Outcome: Progression-free Survival After Initial SPD.
Time Frame: At the time of analysis.
Population: As the study was terminated before the end of recruitment, data was not collected.
Arm/Group | GSK1203486A Group
Number analyzed (Participants) | 0

9. Secondary Outcome: Documentation of Any Toxicity.
Time Frame: During the entire study, up to 2.5 years per patient
Population: As the study was terminated before the end of recruitment, data was not collected.
Arm/Group | GSK1203486A Group
Number analyzed (Participants) | 0

10. Secondary Outcome: Immunogenicity at Defined Time Points.
Time Frame: At 13 defined time points.
Population: As the study was terminated before the end of recruitment, data was not collected.
Arm/Group | GSK1203486A Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All adverse events were collected during the entire study, from Month 0 to early termination date, up to 2.5 years per patient.
Arm/Group | GSK1203486A Group
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1203486A Group (N=5)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1203486A Group (N=5)
Inflammation (Skin and subcutaneous tissue disorders) | 1
Injection site pain (General disorders) | 3
Injection site reaction (General disorders) | 2
Pyrexia (General disorders) | 2
Urinary tract infection (Infections and infestations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (General disorders) | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.